CLINICAL TRIAL: NCT05995977
Title: The Effect of Nursing Interventions Based on Protection Motivation Theory on Drug Adherence and Healthy Lifestyle Behaviors in Patients With Hypertension: A Randomized Controlled Study
Brief Title: Nursing Interventions Based on Protection Motivation Theory in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Handan Altunkan, Principal İnvestigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NecmettinEUHAltunkang9uxfp6y42
Record Dates: First submitted 2023-08-03; First posted 2023-08-16 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hypertension, Public Health; Nursing Staff
Keywords: Nursing, Hypertension, Medication adherence, Protective motivation theory, Healthy lifestyle behaviors.
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: APPLICATION The intervention consists of two components and is planned to last 14 weeks. The first component consists of hypertension education based on CMT. The second component is the sending of regularly delivered KMT-based SMS messages aimed at reminding, encouraging and motivating patients to maintain medication adherence and healthy lifestyle changes.
  Applications made to the intervention group:
  NURSING INITIATIVES
  1. Hypertension Education:
  2. Sending an SMS Message:
  Applications to the control group: No intervention will be applied to the control group by the researcher during the study. Upon the collection of the follow-up test data of the control group, information notes and brochures created within the scope of the research will be given to the patients who request it from this group.
Who Masked: Outcomes Assessor
Masking Description: In order to prevent bias in the evaluation of the data; statistical analyses of the coded data (A and B) in the prepared database were performed by a statistician independent of the researcher. After the statistical analyses of the study and appropriate tables for the results were made and the research report was written, the codings for the control and intervention groups were explained. Thus, statistician and reporting blinding was performed during the research process.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group that applied nursing interventions (Experimental): The intervention consists of two components and is planned to last 14 weeks. The first component consists of hypertension education based on the Protection Motivation Theory. The second component is the sending of regularly delivered Protection Motivation Theory-based SMS messages aimed at reminding, encouraging and motivating patients to maintain medication adherence and healthy lifestyle changes.
  Interventions: Behavioral: Nursing interventions based on protection motivation theory in patients with hypertension
- Individuals who do not apply nursing interventions based on protection motivation theory (No Intervention): Control Group: Individuals who did not apply nursing interventions based on protection motivation theory in patients with hypertension

INTERVENTIONS:
Behavioral: Nursing interventions based on protection motivation theory in patients with hypertension — The intervention consists of two components and is planned to last 14 weeks. The first component consists of hypertension education based on the Protection Motivation Theory. The second component is the sending of regularly delivered Protection Motivation Theory-based SMS messages aimed at reminding, encouraging, and motivating patients to maintain medication adherence and healthy lifestyle changes.
  Arms: Intervention Group that applied nursing interventions

SUMMARY:
Hypertension is a major global public health problem. In order to be successful in hypertension management, patients should receive timely and accurate diagnosis, acquire healthy lifestyle habits, start antihypertensive drug treatment on time, and ensure compliance with treatment. The study was conducted in a pre-test-post-test parallel group randomized controlled design in order to determine the effects of nursing interventions consisting of Rogers' Protection Motivation Terosine-based hypertension education and sending short messages to hypertensive individuals on medication compliance and healthy lifestyle behaviors. The study was conducted in Karaman Province, Family Health Center No. 7 between November 2023 and May 2024. The study group consisted of individuals aged between 40-59 years, with low compliance to treatment, no communication problems in terms of hearing, vision and understanding, using mobile phones, and diagnosed with primary hypertension. The study was conducted with a total of 78 participants, 39 in the intervention group and 39 in the control group, calculated with 95% power. Before starting the study, ethics committee, institution, scale usage permission and written consent were obtained from the participants. Data were collected using Personal Information Form, Antihypertensive Drug Treatment Adherence Scale, Healthy Lifestyle Behaviors Scale, Blood Pressure Monitoring Form at the beginning (T₀), end of the third month (T₁) and end of the sixth month (T₂). Multiple nursing interventions consisting of hypertension education, brochure and 14-week short messages were applied to the intervention group. No intervention was applied to the control group. Measurements were collected by face-to-face interview method. Blinding was applied in terms of statistics expert and reporting. Data analyses in this study were performed using IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA) program. After the applied nursing interventions, a significant difference was found between the total mean score of the Antihypertensive Drug Treatment Adherence Scale, the mean score of the Healthy Lifestyle Behaviors Scale, and systolic blood pressure and diastolic blood pressure values of the intervention and control groups (p<0.05). As a result, applicable, economical interventions combining health education and technology can be recommended as an important tool in health services to reduce the burden of hypertension in society.

DETAILED DESCRIPTION:
In this study, which was conducted to determine the effect of nursing interventions based on the Protection Motivation Theory on medication compliance and healthy lifestyle behaviors in patients with hypertension, 78 adult participants between the ages of 40 and 59 were randomized, and a pre-test was performed using the antihypertensive medication compliance and healthy lifestyle behavior scale and blood pressure measurement. A study will be conducted in a test-post-test controlled design.

Research Universe: The research universe consists of 407 individuals with primary hypertension between the ages of 40-59 registered at the Family Health Center (ASM) No. 7 in Karaman, Turkey.

Sample of the Study: In this study, "G. Sample size was calculated at a 95% confidence level using the "Power-3.1.9.2" program. Özpancar's (2013) study was used for the calculation. The number of samples required for this calculation is 0.05 alpha value for the Mann Whitney U test; The minimum sample size was determined as 70 people in total, 35 for each group (intervention and control), by taking the effect size of 0.90 and the theoretical power of 95%. The 10% loss rate in previous studies was taken into account and it was decided to include a total of 78 participants, 39 in each group. Data Collection Technique and Tools: In the collection of data; Exclusion Criteria Form, Personal Information Form, Antihypertensive Drug Treatment Adherence Scale, Healthy Lifestyle Behaviors Scale, Blood Pressure Monitoring Form, Telephone follow-up form, and short message service follow-up chart were used.

Exclusion Criteria Form: This form was created according to the exclusion and inclusion criteria of the study in order to determine the participants to be included in the study. The form consists of a total of 7 questions (age, education level, primary hypertension diagnosis, a second chronic disease, pregnancy or breastfeeding status, mobile phone use, compliance with antihypertensive drug treatment) and 1 decision to include in the study.

Socio-demographic Information Form: This form was created as a result of literature review. The form consists of a total of 20 questions. 9 determine the socio-demographic characteristics of individuals (age, weight, height, gender, marital status, education status, employment status, monthly income, lifestyle) and are related to hypertension (time of hypertension diagnosis, number of anti-hypertensive drugs used daily, anti-hypertensive drugs used daily). It consists of a total of 20 questions, 11 of which are about duration of hypertensive medication use, regular use of hypertension medication/medicine, place of follow-up treatment, family history of hypertension, diet specific to hypertension, daily tea/coffee consumption, smoking status, alcohol use, regular exercise).

Antihypertensive Medication Adherence Scale: The Turkish validity and reliability of the scale developed by Morisky, Green and Levine was conducted by Demirezen and Nahcivan. The scale includes a total of 9 statements that diagnose medication-taking behavior. The first 8 questions are answered as Yes and No, and yes answers are coded as "1" and no answers as "0". The ninth question has the options "1" never/rarely, "2" occasionally, "3" sometimes, "4" usually, "5" always, and only one option is selected. In scoring, Yes = 0 points and No = 1 points are evaluated in questions 5 and 6, while Yes = 1 and No is evaluated as 0 in other questions. The last question, item 9, is Likert-type and is evaluated between 1-5. The Cronbach's alpha coefficient of the scale was reported as 0.82 in the entire scale. In the study in question, the definitions of compliance and non-compliance with antihypertensive drug treatment were determined according to the 80% cut-off point. In this study, Cronbach's Alpha reliability coefficient was found as 0.674 in the first measurement, 0.797 in the second measurement and 0.748 in the third measurement. An increase in the score in the evaluation of compliance with antihypertensive drug treatment indicates that the individual is "non-compliant". The total scale score varies between '1-13'. Accordingly, individuals who score "1-7" according to the total scale score while participants who scored "8 and above" were defined as non-compliant with treatment.

Healthy Lifestyle Behaviors Scale: Healthy behaviors were collected with the "Healthy Lifestyle Behaviors Scale". The scale was developed by Walker et al. (1987) and revised again in 1996. The scale consists of a total of 52 items and has 6 sub-factors. The sub-groups are spiritual development, health responsibility, physical activity, nutrition, interpersonal relationships and stress management. All items of the scale are positive. The lowest score for the entire scale is 52, the highest score is 208. The rating is in the form of a 4-point Likert. It is accepted as never (1), sometimes (2), often (3), regularly (4). The Cronbach Alpha coefficient of the original scale is 0.94 and the Cronbach Alpha values of the sub-dimensions of the scale vary between 0.79-0.87. The scale was adapted to Turkish by Bahar et al. (2008). In the study in question, the Cronbach alpha reliability coefficient was determined as 0.92. In this study, Cronbach's Alpha reliability coefficient was found to be 0.904 in the first measurement, 0.928 in the second measurement and 0.926 in the third measurement. The scale measures the health-improving behaviors of the individual in relation to a healthy lifestyle.

Blood Pressure Measurement Form: Blood pressure was measured by the researcher with a calibrated mercury-manual sphygmomanometer (Erka Perfect Aneroid/Germany) and a stethoscope.

Data Collection: Hypertensive individuals who agreed to participate in the study were first asked to fill out a pre-test form. The interviews were first conducted face-to-face by the researcher in the training hall of the Family Health Center. After nursing interventions (Hypertension Education Presentation November - December 2023, SMS message sending December 2023 - March 2024), interim measurement data were collected. Post-tests were performed at the end of the sixth month.

Study Variables: Dependent variables: Antihypertensive drug compliance scale mean score, healthy lifestyle behavior scale mean score, systolic and diastolic blood pressure. Independent variables: Nursing interventions based on Protection Motivation Theory Statistical Evaluation of Data: In this study, data analyses were performed using the IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA) program. Descriptive statistics were given as number of units (n), percentage (%), mean (X), standard deviation (SS), median (M), minimum (min) and maximum (max) values. Reliability for scales and their sub-dimensions was examined using Cronbach's Alpha coefficient. Scales with a Cronbach's Alpha coefficient above 0.60 were considered reliable. Skewness and kurtosis values were examined to test whether the data met the assumption of normality. In the decision phase, if the absolute skewness (Skewness) value is below ± 2.0 and the kurtosis value is below 7.0, it is decided that the data is normally distributed. Accordingly, the data in the study was found to be suitable for normal distribution. In the comparison of numerical descriptive characteristics of the patients between groups, independent sample t test was used, and in the comparison of categorical descriptive characteristics between groups, chi-square tests (Pearson chi-square/Fisher exact test) were used. Mixed order analysis of variance (ANOVA) was used in the comparison of variables in the groups according to follow-up times. Bonferroni correction was applied in the comparison of main effects in the analyses. The value of p<0.05 was considered statistically significant. Intention to treat (ITT) analysis was used in the evaluation of the data. ITT is a basic method used in maintaining randomization and preventing bias in case of withdrawal from the study. Since it was not possible to reach 7 individuals who left the research process for the ITT analysis of this study, the post-tests were filled by repeating the answers given by the patients in the pre-tests, and the missing data were completed in this way.

Randomization: Socio-demographic data (age, gender, education level and income level) of hypertensive patients from the 7th FHC where the study was to be conducted were obtained as a list and found to be similar. Therefore, no stratification was applied in the study while determining the sample of the study. In the first stage of the study, hypertensive individuals defined as non-adherent to treatment (scoring "8 and above") were determined by using the antihypertensive drug treatment compliance level scale for individuals registered in the 7th FHC and continuing antihypertensive drug treatment. This process was continued until the specified sample size (n: 78) was reached. Each individual to whom the scale was applied was given a number from 1 to 78 according to the application order and a list was created. In the second stage, participants were assigned to the intervention and control groups from the web page (https://www.random.org/) according to the simple randomization method based on the order in the list created. In this assignment, the assignment of the groups was made by an expert in order to ensure blinding. The flow chart of the control and intervention groups was prepared in accordance with the guidelines specified in CONSORT 2022.

Masking: Patients were invited to the study by the researcher involved in the study and participant registration was carried out until the targeted sample size (78 participants) was reached. During participant registration, the names and contact information of the patients were collected, and it was stated that they would be contacted and called for the process related to the study. When the targeted sample size was reached in the study, participant registration was terminated and a participant list was created. Random selection and assignment were made in the study by a person other than the researcher using the created participant list. Thus, selection bias was controlled in the study. After the groups were determined, the patients were not blinded since their consent would be obtained for the application to be made to them during the intervention process. In this study, a blind technique was applied by hiding who was in the control and intervention groups until the nursing interventions based on KMT started. However, the researcher was not blinded during the intervention period. In order to prevent bias in the evaluation of the data; statistical analyses of the coded data (A and B) in the prepared database were performed by a statistician independent of the researcher. After the statistical analyses of the study and appropriate tables for the results were made and the research report was written, the codings for the control and intervention groups were explained. Thus, statistician and reporting blinding was performed during the research process. Intention to treat analysis (ITT) was applied to prevent attrition bias due to missing data in the outcome/outcome measurements during the study process after randomization. In this way, selection, attrition, statistical and reporting bias were controlled.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been diagnosed with primary hypertension (at least one year)
* Those between the ages of 40 and 59
* Those who use a mobile phone to receive SMS messages sent by the researcher
* Those who are at least literate and can speak Turkish
* Those who have no communication problems in terms of hearing, seeing and understanding
* Those who use antihypertensive medication and who score "8 and above" on the compliance scale and are defined as non-compliant with treatment were decided to be included in the study.

Exclusion Criteria

* Having a second chronic disease
* Those with mental or communication problems
* Those with secondary hypertension (Addison's disease, Renal artery stenosis, Hypo/hyperthyroidism, Parenchymal kidney disease, Cushing's Disease)
* Pregnant or lactating,

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilek CİNGİL, Study Director — dcingil@erbakan.edu.tr
Locations (1):
- Family Health Center No. 7 affiliated with Karaman Provincial Health Directorate, Karaman, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First, 78 (sample number) participants who were not compliant with treatment (scoring "8 and above") were identified using the ASM antihypertensive drug treatment compliance scale. Participants were numbered from one to 78 and a list was created. Based on the order in the list, participants were assigned to the intervention and control groups via the web page (https://www.random.org/) using the simple randomization method. Group assignment was made by an expert to ensure blinding.
Period: Overall Study
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing Interventions Based on Protection Motivation Theory
Started | 39 | 39
Completed | 36 (The study started with 39 participants in the intervention group. Later, 3 people left the study. The patients who left the study stated their reasons for leaving by using expressions such as "my blood pressure is no longer high, I am better, I want to leave your intervention" (n=1). In addition, a total of 2 patients had to be removed from the study by the researcher because the phone numbers they gave could not be reached.) | 35 (The study started with 39 participants in the control group. Later, 4 people left the study. The patients who left the study stated their reasons for leaving by using expressions such as "I am very busy with my work, I can no longer spare time for your work" (n=3), "I cannot walk or diet, I cannot lose weight, I do not want to fill out your survey" (n=1) (Total 4 patients).)
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing Interventions Based on Protection Motivation Theory | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.54 (5.15) | 51.28 (5.12) | 51.41 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 19 | 21 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Scale of Adherence to Antihypertensive Drug Treatment
Description: It was developed by Morisky, Green and Levine. There are a total of 9 statements in the scale that define drug-taking behavior. In the first 8 questions, answers are answered as Yes and No, and yes answers are coded as "1" and no answers as "0". In the ninth question, there are "1" never/rarely, "2" sometimes, "3" sometimes, "4" usually, "5" always and one option is marked. The Cronbach's alpha coefficient of the scale was reported as 0.82 in the whole scale. The total score of the scale varies between '1-13'. In the aforementioned study, the definitions of compatible and incompatible with antihypertensive drug treatment were determined according to the 80% cut-off point. Accordingly, individuals who scored "1-7" according to the total scale score were defined as compatible with the treatment, while participants who scored "8 and above" were defined as non-adherent to the treatment.
Time Frame: Outcomes were assessed at one month (T₀), after the interventions (approximately 3.5 months after baseline) (T₁) and at the end of the sixth month (T₂).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing Interventions Based on Protection Motivation Theory
Number analyzed (Participants) | 39 | 39
score on a scale
  T0 | 9.31 (1.28) | 9.51 (1.21)
  T1 | 7.86 (1.99) | 9.23 (0.84)
  T2 | 8.14 (1.81) | 9.23 (0.84)

2. Primary Outcome: Healthy Lifestyle Behaviors Scale
Description: Scale, Walker et al. (1987) and revised again in 1996 (Walker and Hill-Polerecky 1996). The scale measures health-promoting behaviors associated with an individual's healthy lifestyle. The scale consists of 52 items in total and has 6 sub-factors. Subgroups are spiritual growth, health responsibility, physical activity, nutrition, interpersonal relationships and stress management. The overall score of the scale gives the healthy lifestyle behaviors score. The lowest score for the whole scale is 52, and the highest score is 208. Higher values represent a better result. All items of the scale are positive. The rating is in the form of a 4-point likert. Never (1), sometimes (2), often (3), regularly (4). The Cronbach Alpha coefficient of the original scale is 0.94, and the Cronbach Alpha values of the sub-dimensions of the scale vary between 0.79 and 0.87.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Individuals Who do Not Apply Nursing: Control Group: Individuals who did not apply nursing interventions based on protection motivation theory in patients with hypertension
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing
Number analyzed (Participants) | 39 | 39
score on a scale
  T₀ | 119.90 (11.10) | 119.05 (16.20)
  T₁ | 132.11 (16.76) | 122.23 (12.96)
  T₂ | 131.53 (16.88) | 121.97 (13.08)

3. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure were measured by the researcher using a calibrated mercury-manual sphygmomanometer (sphygmomanometer-Erka Perfect Aneroid/Germany) and stethoscope. Step 1: The patient should rest quietly and comfortably for 5 minutes with his feet flat on the floor and remove the clothes from the arm to be measured. Step 2: Supporting the patient's arm at the level of the right atrium and placing the cuff on the bare arm. Step 3: Palpating the radial artery and inflating the cuff 20-30 mmHg after the loss of the pulse, then relaxing the cuff pressure to 2 mmHg per second and listening for the Korotkoff sounds. Step 4: Determining the first heard sound (Korotkoff 1) as systolic blood pressure, and the last Korotkoff sound as diastolic blood pressure. Step 5: Take two measurements 1-2 minutes apart and take the average of the two readings 6th step: Oral and written presentation of systolic blood pressure and diastolic blood pressure values to the patient
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing Interventions Based on Protection Motivation Theory
Number analyzed (Participants) | 39 | 39
mm Hg
  T₀ | 148.46 (6.50) | 147.82 (6.77)
  T₁ | 140.56 (8.85) | 148.14 (5.95)
  T₂ | 136.81 (11.54) | 148.86 (6.31)

4. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure were measured by the researcher using a calibrated mercury-manual sphygmomanometer (sphygmomanometer-Erka Perfect Aneroid/Germany) and stethoscope. Step 1: The patient should rest quietly and comfortably for 5 minutes with his feet flat on the floor and remove the clothes from the arm to be measured. Step 2: Supporting the patient's arm at the level of the right atrium and placing the cuff on the bare arm. Step 3: Palpating the radial artery and inflating the cuff 20-30 mmHg after the loss of the pulse, then relaxing the cuff pressure to 2 mmHg per second and listening for the Korotkoff sounds. Step 4: Determining the first heard sound (Korotkoff 1) as systolic blood pressure, and the last Korotkoff sound as diastolic blood pressure. Step 5: Take two measurements 1-2 minutes apart and take the average of the two readings 6th step: Oral and written presentation of systolic blood pressure and diastolic blood pressure values to the patient
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing Interventions Based on Protection Motivation Theory
Number analyzed (Participants) | 39 | 39
mm Hg
  T₀ | 93.08 (3.56) | 92.05 (2.74)
  T₁ | 87.78 (4.54) | 90.57 (3.16)
  T₂ | 87.78 (5.79) | 90.43 (2.81)

ADVERSE EVENTS:
Time Frame: Outcomes were assessed at one month (T₀), after the interventions (approximately 3.5 months after baseline) (T₁) and at the end of the sixth month (T₂).
Description: There are no adverse events.
Arm/Group | Intervention Group That Applied Nursing Interventions | Individuals Who do Not Apply Nursing Interventions Based on Protection Motivation Theory
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05995977/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT05995977/SAP_001.pdf
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT05995977/ICF_002.pdf